CLINICAL TRIAL: NCT05062980
Title: A Phase 1/2 Open-Label, Dose-Escalation and Clinical Response Study of Quaratusugene Ozeplasmid in Combination With Pembrolizumab Versus Docetaxel With or Without Ramucirumab in Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: Quaratusugene Ozeplasmid (Reqorsa) in Combination With Pembrolizumab in Previously Treated Non-Small Lung Cancer
Acronym: Acclaim-2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment was slow, due to competition with the many other clinical trials for the same patient population, which led to the decision to end enrollment in the trial.
Sponsor: Genprex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-004
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Tumor suppressor gene 2 (TUSC2); Lipid nanoparticle (LNP); pembrolizumab; Keytruda; Gene therapy; NSCLC; docetaxel; Reqorsa; Acclaim-2; quaratusugene ozeplasmid
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Docetaxel; Ramucirumab

STUDY DESIGN:
Intervention Model Description: Phase 1: 3+3 dose escalation to identify RP2D.
  Phase 2: RP2D expansion cohort followed by parallel randomization in a 2:1 ratio to either investigational arm or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational (Experimental): In Phase 1, the dose expansion portion of Phase 2 and the investigational arm of the randomized portion of Phase 2, patients will receive their assigned dose of quaratusugene ozeplasmid (via intravenous infusion) in combination with a fixed 200 mg dose of pembrolizumab (via intravenous infusion) once in every 21-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Biological: quaratusugene ozeplasmid; Drug: pembrolizumab
- Control (Active Comparator): In the control arm of the randomized portion of Phase 2, patients will receive either 75 mg/m2 docetaxel (via intravenous infusion) with or without 10 mg/kg ramucirumab (via intravenous infusion) -OR- investigator's choice of treatment. The treatment regimen for patients randomized to the control arm, must begin at Cycle 1 Day 1 and continue every 21 days until disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: ramucirumab; Drug: Investigator's Treatment of Choice

INTERVENTIONS:
Biological: quaratusugene ozeplasmid — Quaratusugene ozeplasmid is an experimental non-viral therapy utilizing the TUSC2 gene, designed to target cancer cells by interrupting cell signaling pathways that allow cancer cells to grow, re-establishing pathways that promote cancer cell death and modulating the immune system response against cancer cells.
  Other Names: Reqorsa
  Arms: Investigational
Drug: pembrolizumab — Pembrolizumab is a programmed death receptor-1 (PD-1) blocking antibody indicated for treatment of patients with metastatic NSCLC.
  Other Names: Keytruda
  Arms: Investigational
Drug: docetaxel — Docetaxel is a microtubule inhibitor indicated for locally advanced or metastatic NSCLC after platinum-based chemotherapy failure.
  Other Names: Taxotere
  Arms: Control
Drug: ramucirumab — Ramucirumab is a human vascular endothelial growth factor receptor 2 (VEGFR2) antagonist indicated in combination with docetaxel for treatment of NSCLC with disease progression after platinum-based chemotherapy.
  Other Names: Cyramza
  Arms: Control
Drug: Investigator's Treatment of Choice — Treatment will be administered during 21-day treatment cycles. The investigator's treatment must not include investigational drugs or therapies.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the safety and efficacy of quaratusugene ozeplasmid (Reqorsa), in combination with pembrolizumab in patients with previously treated NSCLC. Quaratusugene ozeplasmid consists of non-viral lipid nanoparticles that encapsulate a DNA plasmid with the TUSC2 tumor suppressor gene, and is a systemic gene therapy.

The study will be conducted in 2 phases, a dose escalation phase (Phase 1) and a safety and efficacy evaluation phase (Phase 2). In Phase 1, patients will be enrolled in sequential cohorts treated with successively higher doses of quaratusugene ozeplasmid in combination with pembrolizumab to determine the recommended Phase 2 dose (RP2D). Phase 2 will be comprised of a dose expansion portion and a randomized portion. In the dose expansion portion, patients will be enrolled and treated with quaratusugene ozeplasmid at the RP2D in combination with pembrolizumab. In the randomized portion, patients will be randomized to receive either the investigational treatment of quaratusugene ozeplasmid at the RP2D in combination with pembrolizumab or a control treatment of either docetaxel +/- ramucirumab or the investigator's treatment of choice.

DETAILED DESCRIPTION:
Acclaim-2 is a Phase 1/2 multicenter, open-label study of quaratusugene ozeplasmid in combination with pembrolizumab in patients with locally advanced or metastatic NSCLC with any PD-L1 TPS and NOT considered refractory to pembrolizumab, as defined by having achieved at least a 3-month clinical benefit to previous pembrolizumab-containing treatment.

The total duration of study for each patient will be dependent upon the safety, tolerability, and efficacy of the study treatment.

The Phase 1 portion of the study will involve a 3+3 dose escalation schema of quaratusugene ozeplasmid up to 0.12 mg/kg in combination with a fixed dose of pembrolizumab (200 mg) administered once via intravenous (IV) infusion during each 21-day treatment cycle. Three quaratusugene ozeplasmid doses will be tested (0.06, 0.09 and 0.12 mg/kg administered on Day 1 of a 21-day treatment cycle).

Phase 2 will involve a dose expansion portion and a randomized portion. In the dose expansion portion 36 patients will be enrolled to better characterize the safety and preliminary efficacy of quaratusugene in combination with pembrolizumab. Patients in the dose expansion portion will receive quaratusugene ozeplasmid at the RP2D determined in Phase 1 in combination with pembrolizumab once in every 21-day treatment cycle. When the PFS rate at 18 weeks has been evaluated for all patients in the dose expansion portion and been shown to meet the criteria for advancement to the randomized portion of Phase 2, the randomized portion of Phase 2 will be initiated. In the randomized portion of Phase 2, 126 patients will be randomized 2:1 to the investigational (quaratusugene ozeplasmid in combination with pembrolizumab) versus control (docetaxel with or without ramucirumab, or investigator's choice of treatment) treatment arms, respectively. Patients will be stratified by NSCLC histology (squamous versus nonsquamous predominant histology) for efficacy analysis purposes. The 84 patients randomized to the investigational arm will receive quaratusugene ozeplasmid, at the RP2D determined in Phase 1, administered in combination with 200 mg pembrolizumab once in every 21-day treatment cycle. The 42 patients randomized to the control arm may either receive docetaxel with or without ramucirumab, or a non-investigational treatment chosen by the investigator.

ELIGIBILITY:
Patients will have their most recent archival tumor biopsy submitted to a central laboratory for IHC analysis.

Inclusion Criteria:

1. Age ≥18 years.
2. Voluntarily signed an informed consent in accordance with institutional policies.
3. Histologically or cytologically documented NSCLC (SQ, NSQ, or mixed (adenosquamous) histology) with locally advanced or metastatic disease. Note: Any level of PD-L1 TPS is allowed.
4. Achieved clinical benefit to prior pembrolizumab or pembrolizumab/platinum-based chemotherapy for at least 3 months and subsequently progressed as confirmed by radiological tumor assessment per RECIST 1.1. Patients receiving pembrolizumab as a single agent must have additional therapy with a platinum-based chemotherapy prior to enrolling, but patients receiving pembrolizumab in combination with a platinum-based chemotherapy should have enrollment in this trial as the next treatment regimen. Chemotherapy is to be limited such that study treatment will be 2nd or 3rd line.
5. For Phase 2, patients must have measurable disease per RECIST 1.1.
6. Patients with genetic alterations with FDA-approved therapy (such as EGFR or anaplastic lymphoma kinase [ALK] mutations) must have disease progression after treatment with appropriate targeted therapy and must be eligible for immunotherapy as determined by the investigator.
7. ECOG performance status score from 0 to 1.
8. Must be ≥28 days beyond major surgical procedures such as thoracotomy, laparotomy, or joint replacement, and must be ≥10 days beyond minor surgical procedures such as biopsy of subcutaneous tumors, pleuroscopy, etc., and must not have evidence of wound dehiscence, active wound infection, or comparable major residual complications of the surgery. Note: Placement of pleural catheter despite being a minor surgical procedure, may be performed <10 days prior to study enrollment.
9. Demonstrate adequate organ function, as determined by the following laboratory values obtained within 21 days prior to enrollment:

   1. Absolute neutrophil count (ANC) ≥1,500/μL,
   2. Platelets ≥ 100,000/μL,
   3. Hemoglobin ≥8.0 g/dL ≥2 weeks without transfusions,
   4. International normalized ratio (INR) or prothrombin time (PT): ≤1.5 × upper limit of normal (ULN) unless the patient is receiving anticoagulant therapy as long as PT is within therapeutic range of intended use of anticoagulants,
   5. Activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT): ≤1.5 × ULN unless the patient is receiving anticoagulant therapy as long as aPTT is within therapeutic range of intended use of anticoagulants,
   6. Creatinine ≤1.5 × ULN OR calculated creatinine clearance (CrCl) ≥60 mL/min for patients with creatinine levels >1.5 × ULN,
   7. Serum total bilirubin ≤1.0 × ULN,
   8. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 × ULN,
   9. Alkaline phosphatase ≤2.5 x ULN.
10. Stable cardiac condition with a left ventricular ejection fraction >40% within ≤21 days prior to enrollment.
11. Asymptomatic brain metastases, must meet ALL of the following criteria (a-d):

    1. No history of seizures in the preceding 6 months,
    2. Definitive treatment must be completed ≥4 weeks prior to enrollment,
    3. Stopped corticosteroid treatments administered because of brain metastases or related symptoms for ≥2 weeks prior to enrollment,
    4. Post-treatment imaging must demonstrate stability or regression of the brain metastases.
12. Female patients of childbearing potential (FOCBP) must have a negative serum pregnancy test at screening (within 7 days of enrollment). Note: Non-childbearing potential is defined as greater than 1 year postmenopausal or surgically sterilized.
13. FOCBP and non-sterile male patients with female partner(s) of childbearing potential must agree to use 2 forms of contraception including 1 highly effective and 1 effective method beginning ≥2 weeks prior to enrollment through 4 months following the last dose of study treatment.
14. Male patients must agree to no sperm donation during study treatment and for an additional 4 months following the last dose of study treatment.

Exclusion Criteria:

1. Unable to tolerate pembrolizumab treatment, leading to early treatment discontinuation or prolonged/frequent dosage modifications as determined by the investigator.
2. Hypersensitivity to docetaxel or polysorbate 80 (Phase 2 only).
3. Patients at risk of tumor lysis syndrome (e.g., renal impairment, hyperuricemia, bulky tumor [Phase 2 randomized portion only]).
4. Received prior systemic chemotherapy or monoclonal antibodies for the treatment of the participant's advanced or metastatic disease within 21 days of study enrollment.
5. Received prior gene therapy.
6. Received any radiotherapy to the skull, spine, thorax, or pelvis within 1 month of study enrollment. Note: Patients are permitted to have received palliative radiotherapy to an extremity provided at least 14 days has elapsed since completion of therapy, provided the patient received no more than 10 radiotherapy fractions and a dose no higher than 30 Gy to that site.
7. Expected to require any other form of antineoplastic therapy while participating in the study.
8. Received a live-virus vaccination within 1 month of enrollment. Seasonal flu vaccines that do not contain live virus are permitted.
9. Has known active, symptomatic CNS metastases and/or carcinomatous meningitis.
10. Active, known, or suspected autoimmune disease.
11. Active systemic viral, bacterial, or fungal infections(s) requiring treatment.
12. Serious concurrent illness or psychological, familial, sociological, geographical, or other condition that, in the opinion of the investigator, would prevent adequate follow-up and compliance with the study protocol.
13. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study enrollment. Inhaled or topical steroids and adrenal replacement doses ≤10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
14. Active concurrent malignancies, i.e., cancers other than NSCLC.
15. Has a second, concurrent, untreated malignancy.
16. History of symptomatic interstitial lung disease or pneumonitis that required oral (PO) or IV glucocorticoids to assist with management. Note: Lymphangitic spread of the NSCLC is not an exclusion criterion.
17. History of myocardial infarction or unstable angina within 6 months prior to enrollment.
18. Presence of pre-existing peripheral neuropathy that is ≥Grade 2 by NCI-CTCAE v5.0 criteria.
19. Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or has a recent history (within the last year) of substance abuse (including alcohol) requiring medical intervention.
20. Known human immunodeficiency virus (HIV) infection or has active hepatitis infection.
21. Female patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) - Phase 1 | First 21-days at each dose level
  RP2D which will be the MTD or if the MTD is not defined by the safety data, the RP2D will be determined based on an integrated assessment of all available clinical safety, PK, and preliminary efficacy data.
Progression-free Survival (PFS) - Phase 2 Dose Expansion | 18 weeks
  PFS rate at 18 weeks after first dose of study treatment. PFS according to RECIST.
Progression-free Survival (PFS) - Phase 2 Randomized | Approximately 8 months
  PFS from randomization to disease progression or death. PFS according to RECIST.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) - Phase 1 | Approximately 8 months
  PFS from first study treatment to disease progression or death. PFS according to RECIST.
Overall Survival (OS) - Phase 1 | Approximately 11 months
  OS from first study treatment to death or discontinuation due to withdrawal of consent.
Pharmacokinetics (PK) - Phase 1 | First 21-day treatment cycle
  Concentrations of quaratusugene ozeplasmid in whole blood samples.
Adverse Events (AEs) - Phase 2 Dose Expansion | Approximately 9 months]
  Number of treatment-related AEs graded according to the NCI-CTCAE.
Progression-free Survival (PFS) - Phase 2 Dose Expansion | Approximately 8 months
  PFS from first study treatment to disease progression or death. PFS according to RECIST.
Overall Response Rate (ORR) - Phase 2 Dose Expansion | Approximately 8 months
  ORR (Complete Response [CR] + Partial Response [PR]) using best overall response from first study treatment to disease progression or death per RECIST compared to baseline tumor measurements.
Overall Survival (OS) - Phase 2 Dose Expansion | Approximately 11 months
  OS from first study treatment to death or discontinuation due to withdrawal of consent.
Pharmacokinetics (PK) - Phase 2 Dose Expansion | First 21-day treatment cycle
  Concentrations of quaratusugene ozeplasmid in whole blood samples.
Overall Response Rate (ORR) - Phase 2 Randomized | Approximately 8 months
  ORR (CR + PR) using best overall response from randomization to disease progression or death per RECIST compared to baseline tumor measurements.
Overall Survival (OS) - Phase 2 Randomized | Approximately 11 months
  OS from randomization to death or discontinuation due to withdrawal of consent.
Disease Control Rate (DCR) - Phase 2 Randomized | Approximately 8 months
  DCR (CR + PR + Stable Disease [SD]) using best overall response from randomization to death or discontinuation due to withdrawal of consent per RECIST compared to baseline tumor measurements.
Adverse Events (AEs) - Phase 2 Randomized | Approximately 9 months
  Number of treatment-related AEs graded according to the NCI-CTCAE.
Pharmacokinetics (PK) - Phase 2 Randomized | First 21-day treatment cycle
  Concentrations of quaratusugene ozeplasmid in whole blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, MD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - Moffitt Cancer Center - Magnolia Campus, Tampa, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Mary Crowley Cancer Research, Dallas, Texas
  - Millennium Oncology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No